CLINICAL TRIAL: NCT06796218
Title: Validity and Reliability of the Arabic Version of De Morton Mobility Index After Abdominal Surgeries
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basant Ashraf Younes Mohamed, Basant Ashraf Younes Mohamed, Cairo University
Other Study IDs: DE Morton index after surgries
Record Dates: First submitted 2025-01-12; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Surgeries; Mobility Limitation; Mobility Difficulty; Abdominal Surgery Patients
Keywords: mobility limitation; mobility difficulty; abdominal surgeries; abdominal surgical approaches
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The study will include106 Egyptian participants of both sexes after abdominal surgeries: The study will include 103 Egyptian participants of both sexes after abdominal surgeries. Their ages range between (60 and 90) years.
  Inclusion criteria:
  1. Patients after abdominal surgeries.
  2. Patients aged between 40 and 60 years.
  3. All patients are able to read and write in Arabic language.
  4. All patients can understand items of the scale.
  5. All patients will follow the given instructions during the assessment.
  Exclusion criteria:
  1. Patients with mental disabilities .
  2. Patients with communication, vision and hearing disorders
  3. Patients who are not co-operative .
  4. patients who are contraindicated to mobilize due to medical reasons.
  5. patients who are isolated due to infection.

SUMMARY:
PURPOSE: To determine validity and reliability of translated Arabic version of the De Morton Mobility index for mobility assessment in patients after abdominal surgeries.

BACKGROUND:

Major abdominal surgery has a high morbidity and Mortality rate, and the risk of surgical complications is higher than for equivalent elective operations. those receiving emergency laparotomy are in a condition of physiological derangement driven by inflammation that has already occurred prior to surgery, in contrast to those undergoing elective abdominal operations. early mobility and exercise play an important role in postoperative treatment following abdominal surgery and are related with reduced postoperative fitness loss and fewer postoperative complications in individuals undergoing elective surgery. reduced mobility is a primary factor of lower quality of life and decreased social participation. reduced mobility is particularly common in older hospitalized patients, and it leads to an increased risk of falls, longer hospitalizations, more severe impairment and morbidity, and higher mortality rates. To manage elderly patients' mobility function, a reliable and valid mobility assessment tool is required. Performance-based examinations are commonly used to measure the mobility of elderly individuals. The De Morton Mobility Index (DEMMI) was established and validated exclusively for older patients hospitalized in the ward. The DEMMI provides clinicians and researchers with a valid interval-level method for accurately measuring and monitoring mobility levels of acute medical patients. It has been validated also in sub acute hospital and community settings. A DEMMI score of <40 indicates an independent risk of serious postoperative complications. A low DEMMI score suggested impaired mobilization, and prior research of patients following abdominal surgery discovered that delayed mobilization was related with postoperative pulmonary complications.

HYPOTHESES: It will be hypothesized that: Arabic version of the De Morton Mobility Index may be valid and reliable in patients after abdominal surgeries.

RESEARCH QUESTION: Is The Arabic version of the De Morton Mobility index valid and reliable for mobility assessment in patients after abdominal surgeries?

DETAILED DESCRIPTION:
This study will be designed to assess the validity and reliability of the Arabic version of De Morton mobility index in patients after abdominal surgeries.

Study Design: This study is designed as a cross-sectional study. Subjects: The study will include 106 Egyptian participants of both sexes after abdominal surgeries. Their ages range between (40 and 60) years .They will be selected randomly from: Mansoura International Hospital .

Material: Data will be collected mainly from Mansoura Hospitals through the use of The Arabic version of De Morton Mobility Index.

study scale and its scoring: The De Morton Mobility Index (DEMMI) is a 15-item clinician-rated performance-based measure of mobility in older adults. The DEMMI has minimal equipment requirements and the scale protocol and scoring system fit onto one page. Only a bed or plinth, armchair (seat height 45 cm) and pen are required to conduct the test.

The 15 tasks will be given in order of difficulty, beginning with bed (3 items), then chair (3 items), static balance (4 items), walking (2 items), and dynamic balance (3 items). The overall score runs from 0 to 100, with 0 representing severely limited physical mobility and 100 indicating independent mobility. Any competent healthcare provider can administer the DEMMI with minimum equipment.

Methods: This study will follow the guidelines of Sousa in translation. Step 1: Forward translation (Initial translation) Step 2: Synthesis of translation Step 3: Backward translation Step 4: Expert review Step 5: Test of pre-final testing Step 6: Authentication Psychometric properties: The final Arabic version of DE Morton Mobility Index will be assessed with regard to the validity and reliability using psychometric tests.

The scores will be administered twice to ensure test/retest reliability. The first score was obtained immediately following the procedure, and the second one week later.

ELIGIBILITY:
Inclusion Criteria:

1. Patients after abdominal surgeries.
2. Patients aged between 40 and 60 years.
3. All patients are able to read and write in Arabic language.
4. All patients can understand items of the scale.
5. All patients will follow the given instructions during the assessment

Exclusion Criteria:

1. Patients with mental disabilities .
2. Patients with communication, vision and hearing disorders
3. Patients who are not co-operative .
4. patients who are contraindicated to mobilize due to medical reasons.
5. patients who are isolated due to infection.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include 106 Egyptian participants of both sexes after abdominal surgeries. Their ages range between (40 and 60) years .They will be selected randomly from:
  • Mansoura International Hospital .
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
validity of de morton mobility index | 3 months from September,2024 to December, 2024
  De morton mobility index is a scale for mobility assessment. it's score ranges from 0 (the minimum) to 19 the maximum(which is the best ). Clarity index and expert proportion of the clearance were used to test( face validity).
  Index of content validity (CVI), scale content validity indices (S-CVI) and expert proportion of relevance were used to test the (content validity).
reliability of De morton mobility index | 3 months from September, 2024 to December, 2024
  Cronbach's alpha will be used to measure the internal consistency reliability. Test-retest reliability will be measured using intraclass correlation coefficient (ICC). The level of significance for all statistical tests will be set at p < 0.05. the study includes 103 participants the lowest score (minimum )for this scale is 0 (worse outcome) the highest score (maximum) for this scale is 19 (interpreted as better outcome) the conversion table's scores ranged from (0 to 100) DEMMI is the abbreviation of De Morton Mobility Index.

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Othman, professor, Study Chair — faculty of physical therapy, department of surgery, cairo university.; Karim I Saafan, Professor, Study Chair — faculty of physical therapy, department of surgery, cairo university.; Amr A Abouzid, professor, Study Chair — Faculty of Medicine, Mansoura University; Basant A younes, B.Sc.of PT, Principal Investigator — B.Sc., Faculty of Physical Therapy, Department of PT for Surgery, Delta University
Locations (1):
- El-Mansoura international hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: De Morton, N. A., Davidson, M., & Keating, J. L. (2008). The de Morton Mobility Index (DEMMI): An essential health index for an ageing world. Health and Quality of Life Outcomes, 6 — https://hqlo.biomedcentral.com/articles/10.1186/1477-7525-6-63